CLINICAL TRIAL: NCT00037960
Title: Automated Constraint-Induced Therapy for Restoring Movement After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2480T
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2002-05

CONDITIONS: Cerebrovascular Accident
Keywords: Constrained Induced; CI therapy; CVA; Strokes
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

INTERVENTIONS:
Procedure: Constrained Induced Therapy

SUMMARY:
We propose to develop and evaluate a workstation that significantly enhances the application of Constraint-Induced (CI) Therapy by automating and instrumenting several of the tasks currently used in the shaping training. The motivation for development of such a device is as follows: 1) Patients could receive CI therapy at home without the need for constant supervision from a therapist. Many veterans do not have the resources to travel to their local VAMC for the two or three week period required for the treatment. A home-based device would expand the pool of veterans who could receive CI therapy. 2) For subjects who were able to receive CI therapy in the clinic, this device would facilitate an effective post-treatment home-practice program. 3) Currently, patients are treated on a one-on-one basis in the clinic. This device could allow one therapist to treat 3 or 4 patients at one time, thereby substantially reducing the cost of the therapy. 4) This workstation would provide clear and comprehensive quantification of the progress of the treatment. This could indicate on which tasks the patient was progressing most and least rapidly, and would therefore enable effective modifications of the treatment plan while treatment was in progress.

The hypothesis is that the positive outcomes of CI therapy can be achieved, and possibly enhanced, if the shaping training component is performed in a workstation that guides, motivates and records exercise of the more-affected limb. In the first 18 months, the workstation will be designed and fabricated. To expedite the design, we will rely on simple modifications to "off the shelf" components. In the last 18 months, a controlled, randomized, clinical trial will compare the effectiveness of automated CI therapy programs with standard CI therapy. The standard CI therapy group would receive shaping training in a clinical setting, one-on-one with a therapist. The clinic-based automated CI therapy group would perform the shaping training in the workstation, in a clinical setting and with minimal supervision. The home-based automated CI therapy group would perform the shaping training at home in the workstation, and with no direct supervision. All other aspects of the three treatment programs will be identical. At the end of this 3-year project, a device will have been designed, built and evaluated that could significantly enhance the application of CI therapy for chronic stroke patients.

DETAILED DESCRIPTION:
Cerebrovascular accident (CVA) is the leading cause of disability in the United States. CVAs are a particular problem for the VA because of the large population of World War II and Korean War veterans who are now in the age range where CVAs are most frequent; in fiscal year 1997 the national VA system had 22,000 admissions for an acute CVA. The consequent motor deficits that veterans sustain result in very large costs to the VA and the Federal Government. The reduction of CVA-related disability thus represents a high VA and national health care priority.

Constraint-Induced (CI) therapy is one of the few techniques that has been proven with controlled, randomized studies to substantially reduce the incapacitating motor deficit of the more-affected upper extremity of patients with mild to moderately severe chronic strokes. The procedures of CI therapy are relatively simple and are deemed effective because they produce transfer of increased extremity use to the activities of daily living in the real world environment. The therapy involves promoting use of the more-affected upper extremity for 90% of waking hours by constraining the less-affected extremity for two or three consecutive weeks with a resting hand splint and sling or other device which prevents movement of the hand and wrist for activities of daily living. The patients receive a type of training termed "shaping" for 7 hours/day (with rest intervals) for all weekdays during this period (massed practice).

We propose to develop and evaluate a workstation that significantly enhances the application of CI therapy by automating and instrumenting several of the tasks currently used in the shaping training. The motivation for development of such a device is as follows: 1) Patients could receive CI therapy at home without the need for constant supervision from a therapist. Many veterans do not have the resources to travel to their local VAMC for the two or three week period required for the treatment. A home-based device would expand the pool of veterans who could receive CI therapy. 2) For subjects who were able to receive CI therapy in the clinic, this device would facilitate an effective post-treatment home-practice program. 3) Currently, patients are treated on a one-on-one basis in the clinic. This device could allow one therapist to treat 3 or 4 patients at one time, thereby substantially reducing the cost of the therapy. 4) This workstation would provide clear and comprehensive quantification of the progress of the treatment. This could indicate on which tasks the patient was progressing most and least rapidly, and would therefore enable effective modifications of the treatment plan while treatment was in progress.

The hypothesis is that the positive outcomes of CI therapy can be achieved, and possibly enhanced, if the shaping training component is performed in a workstation that guides, motivates and records exercise of the more-affected limb. In the first 18 months, the workstation will be designed and fabricated. To expedite the design, we will rely on simple modifications to "off the shelf" components. In the last 18 months, a controlled, randomized, clinical trial will compare the effectiveness of automated CI therapy programs with standard CI therapy. The standard CI therapy group would receive shaping training in a clinical setting, one-on-one with a therapist. The clinic-based automated CI therapy group would perform the shaping training in the workstation, in a clinical setting and with minimal supervision. The home-based automated CI therapy group would perform the shaping training at home in the workstation, and with no direct supervision. All other aspects of the three treatment programs will be identical. At the end of this 3-year project, a device will have been designed, built and evaluated that could significantly enhance the application of CI therapy for chronic stroke patients.

ELIGIBILITY:
Stroke patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wolff, Ph.D. Special Assistant to the Director — Program Analysis and Review Section (PARS), VA Rehabilitation Research & Development Service; Danielle Kerkovitch, Ph.D. — Program Analysis and Review Section (PARS), VA Rehabilitation Research and Development Service; Edward Taub, Ph.D. — University of Alabama at Birmingham
Locations (1):
- VA Medical Center, Palo Alto, California, United States